CLINICAL TRIAL: NCT06146010
Title: Deutsches Meningeosis Neoplastica Register
Brief Title: Non Interventional German Leptomeningeal Disease Register
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: Meningeosis Register
Record Dates: First submitted 2023-11-06; First posted 2023-11-24 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-11

CONDITIONS: Meningeal Neoplasms; Leptomeningeal Disease
Keywords: Meningeosis Neoplastica
MeSH Terms: conditions — Meningeal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- german leptomeningeal disease register: The aim of the leptomeningeal disease register is to establish an internet-based cancer register in which patients with leptomeningeal disease are recorded at the time of diagnosis and after appropriate information and consent to data collection. Due to the rapid progression of the disease and potential rapid deterioration, inclusion must take place at the time of diagnosis. The course of the disease in individual patients is then documented retrospectively on the basis of routine clinical care data for the entire duration of the study or until the death of the participating patients.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Once the patient or their legal guardian has given their written consent, a patient is included in the leptomeningeal disease register. Due to the rapid course of the disease and potential rapid deterioration, the documentation of the course of the disease of the individual patients is to be carried out retrospectively from the data recorded during the course of the clinical routine for the entire duration of the study or until the death of the participating patients after the written consent of the patients. The registry's data sources are the diagnostic findings made at the center and doctors' letters from routine clinical practice. The participating centers carry out the assessment of the participants' performance status so that the patients do not have to complete any study-related questionnaires.

SUMMARY:
The planned multicenter register is intended to create a database in the form of a cancer register on the incidence and course of disease in Germany of leptomeningeal disease, the therapeutic measures administered in the real world and the complications.

DETAILED DESCRIPTION:
This register is multicenter project in Germany. All patients eligible for this register are informed in detail about the register verbally and in writing by the treating and documenting physicians. The written declaration of consent is attached to the patient information form. A patient will only be included in this register once the written declaration of consent has been provided by the patient or their legal guardian. Patient information and the obtaining of consent forms are carried out by the treating medical colleagues.

The register's data sources are the diagnostic findings made at the center and doctors' letters from routine clinical practice. The participating sites carry out the assessment of the participants' performance status so that the patients do not have to complete any study-related questionnaires. There is no intervention in this trial: neither changes to medication nor interventions on the patient themselves are carried out. Invasive measures are not carried out and there is no health risk associated with participation. Within the project, only the occurrence and severity of a neoplastic central nervous system infestation as well as the respective therapeutic measures and their results are documented.

Planned start of register: Quarter 1 2024 Expected end of register: Quarter 4 2029. Once the patient or their legal guardian has given written consent, a patient will be included in the German Meningeosis neoplastica Register. Due to the rapid course of the disease and potential rapid deterioration, the documentation of the course of the disease of the individual patients is to be carried out retrospectively from the clinical routine data recorded during the course of the study for the entire duration of the study or until the death of the participating patients after the written consent of the patients.

There is no minimum or maximum number of patients to be enrolled in this trial. Only descriptive analyses are planned for the data documented in the register.

In accordance with the Declaration of Helsinki/Tokyo/Venice/Hong Kong, all patients have the right to discontinue their participation in the register at any time and without giving reasons, without losing their right to further treatment or experiencing disadvantages of any other kind as a result. The data is pseudonymized and can be decrypted using the separately maintained key list. If a patient subsequently withdraws their consent to participate and requests that the data be deleted, this can be done after decryption using the key list. As this is a pure register study without study intervention, there are no plans to discontinue the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with leptomeningeal disease
* Written consent of the patient or legal guardian.
* Capacity to give consent or legal guardianship
* Age ≥ 18 years

Exclusion Criteria:

* Lack of informed consent from the patient
* Lack of capacity to consent on the part of the person concerned or lack of legal guardianship
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The majority of patients observed are capable of giving consent. However, tumors of the central nervous system can lead to a psychosyndrome that restricts the patient's ability to give consent. Nevertheless, it is important to document and evaluate the course of the disease and the effects of the therapies administered, especially in these patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival depending on the treatment modalities | through study completion, an average of 1 year
  Only descriptive analyses are planned for the data documented in the register. Absolute and percentage frequencies including two-sided 95% confidence intervals are determined for the frequency of use of certain treatment regimens.
Overall survival depending on the treatment modalities | through study completion, an average of 1 year
  Only descriptive analyses are planned for the data documented in the register. Absolute and percentage frequencies including two-sided 95% confidence intervals are determined for the frequency of use of certain treatment regimens.

SECONDARY OUTCOMES:
Frequency of adverse events during the course of the disease. | through study completion, an average of 1 year
  With regard to the effect of the documented therapies, absolute and percentage frequencies for treatment response including two-sided 95% confidence intervals are determined. For censored data (OS, PFS), survival probabilities including two-sided 95% confidence intervals are determined using the Kaplan Meier method. Events are collected retrospectively and presented using line listings and frequency tables.

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - Universitätsklinikum Bonn Klinik und Poliklinik für Neurologie, Bonn
  - Universitätsmedizin Mannheim Universitätsklinikum Mannheim GmbH Klinik für Neurologie, Mannheim
  - Klinikum rechts der Isar | Technische Universität München; Klinik für Radioonkologie und Strahlentherapie, München
  - Diakonie Klinikum GmbH • Jung-Stilling-KrankenhausAbteilung Neurochirurgie, Siegen
  - University Hospital Tübingen, Neurooncology, Tübingen
  - Universitätsklinikum Ulm; Klinik für Innere Medizin III, Ulm

IPD SHARING:
Plan to Share IPD: No